CLINICAL TRIAL: NCT03843463
Title: Escitalopram and Language Intervention for Subacute Aphasia (ELISA)
Brief Title: Escitalopram and Language Intervention for Subacute Aphasia
Acronym: ELISA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of South Carolina (Other); Medical University of South Carolina (Other); University of California, Irvine (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00268564; P50DC014664 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naming Treatment + Escitalopram (Experimental): 10 mg escitalopram daily for three months (escalating from 5 mg per day for the first week and tapering to 5 mg per day for the last two weeks)
  Interventions: Drug: Escitalopram 10mg; Behavioral: Computer-delivered naming treatment
- Naming Treatment + Placebo (Placebo Comparator): 10 mg placebo daily for three months
  Interventions: Drug: Placebo; Behavioral: Computer-delivered naming treatment

INTERVENTIONS:
Drug: Escitalopram 10mg — Escitalopram tablet
  Other Names: Lexapro
  Arms: Naming Treatment + Escitalopram
Drug: Placebo — Sugar pill manufactured to mimic escitalopram 10 mg tablet
  Other Names: Placebo (for Escitalopram)
  Arms: Naming Treatment + Placebo
Behavioral: Computer-delivered naming treatment — 15 45-minute sessions of computer-delivered naming treatment beginning two months following stroke
  Other Names: Computer-delivered naming treatment (CoDeNT)

SUMMARY:
In this project, the investigators will investigate the effects of a selective serotonin reuptake inhibitor (SSRI), escitalopram, on augmenting language therapy effectiveness, as measured by naming untrained pictures and describing pictures, in individuals with aphasia in the acute and subacute post stroke period (i.e., within three months post stroke).

DETAILED DESCRIPTION:
In this project, the investigators will investigate the effects of a selective serotonin reuptake inhibitor (SSRI), escitalopram, on augmenting language therapy effectiveness, as measured by naming untrained pictures and describing pictures, in individuals with aphasia in the acute and subacute post stroke period (i.e., within three months post stroke). There has been no previous randomized controlled trial (RCT) to evaluate the effect of daily SSRI in the first three months after stroke on improvement of language in people undergoing aphasia treatment. It is plausible that SSRIs, which elevate synaptic serotonin, might enhance recovery by augmenting synaptic plasticity.

The investigators propose to conduct a Phase 2 multi-center, randomized, double blind, placebo-controlled trial of escitalopram for augmenting language intervention in subacute stroke. The investigators hypothesize that daily escitalopram for 90 days after stroke results in greater improvement (compared to placebo) in naming untrained pictures, as well as greater increase in content of picture description and greater improvement in morphosyntactic production, when combined with speech and language treatment (SALT). A second aim is to evaluate the mechanisms of language recovery in individuals who receive active medical treatment and those who receive placebo, using resting state functional magnetic resonance imaging (rsfMRI) and genetic testing. The investigators hypothesize that greater improvement in language is associated with increased connectivity within the left hemisphere language network on rsfMRI in participants who receive escitalopram than in those who receive placebo, independently of improvement in depression. The investigators also hypothesize that the effects are greatest in individuals with val/val allele of brain-derived neurotrophic factor (BDNF) - (consistent with previous studies showing a greater response to treatment and greater neuroplasticity in people with the val/val allele than those with one or more met alleles.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have sustained an acute ischemic left hemisphere stroke.
* Participants must be fluent speakers of English by self-report.
* Participants must be capable of giving informed consent or indicating a legally authorized representative to provide informed consent.
* Participants must be age 18 or older.
* Participants must be within 5 days of onset of stroke.
* Participants must be pre-morbidly right-handed by self-report.
* Participants must have an aphasia diagnosis as confirmed by the Western Aphasia Battery-Revised (Aphasia Quotient < 93.8).

Exclusion Criteria:

* Previous neurological disease affecting the brain including previous symptomatic stroke
* Diagnosis of schizophrenia, autism, or other psychiatric or neurological condition that affects naming/language
* A history of additional risk factors for torsades de pointes (TdP; e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Current severe depression, defined as a score of > 15 on the Patient Health Questionnaire (PHQ-9)
* Uncorrected visual loss or hearing loss by self-report
* Use of any medication approved by the FDA for treatment of depression at the time of stroke onset
* Concomitant use of any monoamine oxidase inhibitors (MAOIs) or pimozide, or other drugs that prolong the QT/QTc interval, triptans (and other 5-Hydroxytryptamine Receptor Agonists), or other contraindications to escitalopram that may be identified.
* A QTc greater than 450 milliseconds on electrocardiogram or evidence of hyponatremia (Na < 130) at baseline
* Pregnancy at the time of stroke or planning to become pregnant during the study term.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Change in Philadelphia Naming Test short-form accuracy score | Baseline, 1 week after computer-delivered naming treatment
  Number of correctly named items of 30 total items on the computerized picture naming assessment. Scores ranges from 0 to 30 with higher scores meaning better naming ability.

SECONDARY OUTCOMES:
Language production as assessed by lexical features of discourse in "Cookie Theft" picture description | Baseline, 5 weeks after computer-delivered naming treatment
  Lexical features, meaning carrying units of language (morphemes), will be counted for each Cookie Theft picture description. There is no maximum number of meaning carrying units, but norms are available to assist in the interpretation of this performance.
Language production as assessed by content units included in picture description of "Cookie Theft" | Baseline, 5 weeks after computer-delivered naming treatment
  Content units are based on a standard scoring template of commonly identified concepts (nouns and verbs) in the left and right regions of the "Cookie Theft" picture. Participants either include or fail to include 30 concepts on the left side of the picture and 23 concepts on the right side of the picture. A ratio of included left content units to included right content units then can be calculated and interpreted as a measure of hemispatial attention.
Language production as assessed by rate of syllables per content unit produced in "Cookie Theft" picture description | Baseline, 5 weeks after computer-delivered naming treatment
  Syllables included in the picture description are counted. Content units are based on a standard scoring template of commonly identified concepts (nouns and verbs) in the left and right regions of the "Cookie Theft" picture. Participants either include or fail to include 30 concepts on the left side of the picture and 23 concepts on the right side of the picture. The average rate of syllables per content unit produced can then be calculated and interpreted as a measure of efficiency in producing relevant information in the task.
Depression as assessed by Patient Health Questionnaire (PHQ-9) | Baseline, 1 week after computer-delivered naming treatment
  9 item scale scored 0-3 for each item. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression. PHQ-9 >15 or suicidal ideation suggest depression sufficient for exclusion or removal from study.
Language production as assessed by Morphosyntactic Generation (MorGen) Test | Baseline, 1 week after computer-delivered naming treatment
  60 item assessment of word morphology (e.g., plurals, possessives) and modifiers (e.g., number, size, color). Each item is scored based on produced accurate descriptors of an image relative to a second reference image (e.g., patients see two trees, one larger than the other, and the phrase "little tree" is elicited). Patients are scored for objects correctly named (nouns) out of 60, instances of correct use of plural marker out of 31, instances of correct use of numbers out of 8, instances of correct modifiers denoting size out of 16, instances of correct modifiers denoting color out of 19, instances of correct modifiers denoting possessive markers out of 17, and instances of correctly named possessing individuals (proper names provided on screen) out of 17. These scores can then be interpreted separately or averaged to interpret a broad morphosyntactic accuracy score.
Stroke severity as assessed by NIH Stroke Scale (NIHSS) | Baseline, 5 weeks after computer-delivered naming treatment, 20 weeks after computer-delivered naming treatment
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patient's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items.
Post-stroke level of disability as assessed by modified Rankin Scale (mRS) | Baseline, 1 week after computer-delivered naming treatment
  The mRS is a 6-level scale from "0-No symptoms" to "6-dead" used to evaluate the degree of disability in patients who have suffered a stroke.
Stroke paresis severity as assessed by right hand strength | Baseline, 1 week after computer-delivered naming treatment
  Right hand strength assessment by dynamometer
Stroke paresis severity as assessed by right hand dexterity | Baseline, 1 week after computer-delivered naming treatment
  Right hand dexterity assessment by 9 peg board test
Change in new vocabulary items as assessed by lexical diversity included in story retelling of "Cinderella" | Baseline, 1 week after computer-delivered naming treatment
  Change in new vocabulary items will be counted for each noun, verb, and adjective in the Cinderella retelling. There is no maximum measure of lexical diversity, but norms are available to assist in the interpretation of this performance.
Change in incidence of new vocabulary items as assessed by lexical diversity included in story retelling of "Cinderella" | Baseline, 1 week after computer-delivered naming treatment
  Change in incidence of each new item will be counted for each noun, verb, and adjective in the Cinderella retelling. There is no maximum measure of lexical diversity, but norms are available to assist in the interpretation of this performance.
Change in language production as assessed by speech errors produced during the story retelling of "Cinderella" | Baseline, 1 week after computer-delivered naming treatment
  Change in number of errors will be counted after each retelling is recorded
Change in Language production as assessed by speech pauses produced during the story retelling of "Cinderella" | Baseline, 1 week after computer-delivered naming treatment
  Change in pauses will be counted after each retelling is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Argye Hillis-Trupe, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhogal SK, Teasell R, Speechley M. Intensity of aphasia therapy, impact on recovery. Stroke. 2003 Apr;34(4):987-93. doi: 10.1161/01.STR.0000062343.64383.D0. Epub 2003 Mar 20. PMID 12649521
- [Background] Brady MC, Kelly H, Godwin J, Enderby P, Campbell P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2016 Jun 1;2016(6):CD000425. doi: 10.1002/14651858.CD000425.pub4. PMID 27245310
- [Background] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670
- [Background] FOCUS Trial Collaboration. Effects of fluoxetine on functional outcomes after acute stroke (FOCUS): a pragmatic, double-blind, randomised, controlled trial. Lancet. 2019 Jan 19;393(10168):265-274. doi: 10.1016/S0140-6736(18)32823-X. Epub 2018 Dec 5. PMID 30528472
- [Background] Doron R, Lotan D, Versano Z, Benatav L, Franko M, Armoza S, Kately N, Rehavi M. Escitalopram or novel herbal mixture treatments during or following exposure to stress reduce anxiety-like behavior through corticosterone and BDNF modifications. PLoS One. 2014 Apr 1;9(4):e91455. doi: 10.1371/journal.pone.0091455. eCollection 2014. PMID 24690945
- [Background] Enderby P, Broeckx J, Hospers W, Schildermans F, Deberdt W. Effect of piracetam on recovery and rehabilitation after stroke: a double-blind, placebo-controlled study. Clin Neuropharmacol. 1994 Aug;17(4):320-31. doi: 10.1097/00002826-199408000-00003. PMID 9316679
- [Background] Fridriksson J, Elm J, Stark BC, Basilakos A, Rorden C, Sen S, George MS, Gottfried M, Bonilha L. BDNF genotype and tDCS interaction in aphasia treatment. Brain Stimul. 2018 Nov-Dec;11(6):1276-1281. doi: 10.1016/j.brs.2018.08.009. Epub 2018 Aug 18. PMID 30150003
- [Background] Gu SC, Wang CD. Early Selective Serotonin Reuptake Inhibitors for Recovery after Stroke: A Meta-Analysis and Trial Sequential Analysis. J Stroke Cerebrovasc Dis. 2018 May;27(5):1178-1189. doi: 10.1016/j.jstrokecerebrovasdis.2017.11.031. Epub 2017 Dec 21. PMID 29276014
- [Background] Hayasaka Y, Purgato M, Magni LR, Ogawa Y, Takeshima N, Cipriani A, Barbui C, Leucht S, Furukawa TA. Dose equivalents of antidepressants: Evidence-based recommendations from randomized controlled trials. J Affect Disord. 2015 Jul 15;180:179-84. doi: 10.1016/j.jad.2015.03.021. Epub 2015 Mar 31. PMID 25911132
- [Background] Hillis AE. The 'standard' for poststroke aphasia recovery. Stroke. 2010 Jul;41(7):1316-7. doi: 10.1161/STROKEAHA.110.585364. Epub 2010 Jun 10. No abstract available. PMID 20538691
- [Background] Hillis AE, Beh YY, Sebastian R, Breining B, Tippett DC, Wright A, Saxena S, Rorden C, Bonilha L, Basilakos A, Yourganov G, Fridriksson J. Predicting recovery in acute poststroke aphasia. Ann Neurol. 2018 Mar;83(3):612-622. doi: 10.1002/ana.25184. Epub 2018 Mar 10. PMID 29451321
- [Background] Hillis AE, Tippett DC. Stroke Recovery: Surprising Influences and Residual Consequences. Adv Med. 2014;2014:378263. doi: 10.1155/2014/378263. PMID 25844378
- [Background] Huber W, Willmes K, Poeck K, Van Vleymen B, Deberdt W. Piracetam as an adjuvant to language therapy for aphasia: a randomized double-blind placebo-controlled pilot study. Arch Phys Med Rehabil. 1997 Mar;78(3):245-50. doi: 10.1016/s0003-9993(97)90028-9. PMID 9084344
- [Background] Jorge RE, Acion L, Moser D, Adams HP Jr, Robinson RG. Escitalopram and enhancement of cognitive recovery following stroke. Arch Gen Psychiatry. 2010 Feb;67(2):187-96. doi: 10.1001/archgenpsychiatry.2009.185. PMID 20124118
- [Background] Kraglund KL, Mortensen JK, Damsbo AG, Modrau B, Simonsen SA, Iversen HK, Madsen M, Grove EL, Johnsen SP, Andersen G. Neuroregeneration and Vascular Protection by Citalopram in Acute Ischemic Stroke (TALOS). Stroke. 2018 Nov;49(11):2568-2576. doi: 10.1161/STROKEAHA.117.020067. PMID 30355209
- [Background] Kurland J, Pulvermuller F, Silva N, Burke K, Andrianopoulos M. Constrained versus unconstrained intensive language therapy in two individuals with chronic, moderate-to-severe aphasia and apraxia of speech: behavioral and fMRI outcomes. Am J Speech Lang Pathol. 2012 May;21(2):S65-87. doi: 10.1044/1058-0360(2012/11-0113). Epub 2012 Jan 31. PMID 22294409
- [Background] Lam RW. Antidepressants and QTc prolongation. J Psychiatry Neurosci. 2013 Mar;38(2):E5-6. doi: 10.1503/jpn.120256. No abstract available. PMID 23422053
- [Background] Lazar RM, Minzer B, Antoniello D, Festa JR, Krakauer JW, Marshall RS. Improvement in aphasia scores after stroke is well predicted by initial severity. Stroke. 2010 Jul;41(7):1485-8. doi: 10.1161/STROKEAHA.109.577338. Epub 2010 Jun 10. PMID 20538700
- [Background] Marangolo P, Fiori V, Sabatini U, De Pasquale G, Razzano C, Caltagirone C, Gili T. Bilateral Transcranial Direct Current Stimulation Language Treatment Enhances Functional Connectivity in the Left Hemisphere: Preliminary Data from Aphasia. J Cogn Neurosci. 2016 May;28(5):724-38. doi: 10.1162/jocn_a_00927. Epub 2016 Jan 25. PMID 26807842
- [Background] Mead GE, Hsieh CF, Lee R, Kutlubaev MA, Claxton A, Hankey GJ, Hackett ML. Selective serotonin reuptake inhibitors (SSRIs) for stroke recovery. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD009286. doi: 10.1002/14651858.CD009286.pub2. PMID 23152272
- [Background] Pan XL, Chen HF, Cheng X, Hu CC, Wang JW, Fu YM, Kong HM, Shao HJ. Effects of Paroxetine on Motor and Cognitive Function Recovery in Patients with Non-Depressed Ischemic Stroke: An Open Randomized Controlled Study. Brain Impairment. 2018 May:1-7.
- [Background] Saeterdal I, Pike E, Ringerike T, Gjertsen MK. Efficacy and Safety for the Newer Antidepressants in Adults [Internet]. Oslo, Norway: Knowledge Centre for the Health Services at The Norwegian Institute of Public Health (NIPH); 2007 Jun. Report from Norwegian Knowledge Centre for the Health Services (NOKC) No. 17-2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK464856/ PMID 29320072
- [Background] Sanchez C, Reines EH, Montgomery SA. A comparative review of escitalopram, paroxetine, and sertraline: Are they all alike? Int Clin Psychopharmacol. 2014 Jul;29(4):185-96. doi: 10.1097/YIC.0000000000000023. PMID 24424469
- [Background] Sebastian R, Saxena S, Tsapkini K, Faria AV, Long C, Wright A, Davis C, Tippett DC, Mourdoukoutas AP, Bikson M, Celnik P, Hillis AE. Cerebellar tDCS: A Novel Approach to Augment Language Treatment Post-stroke. Front Hum Neurosci. 2017 Jan 12;10:695. doi: 10.3389/fnhum.2016.00695. eCollection 2016. PMID 28127284
- [Background] Wang C, Zhang Y, Liu B, Long H, Yu C, Jiang T. Dosage effects of BDNF Val66Met polymorphism on cortical surface area and functional connectivity. J Neurosci. 2014 Feb 12;34(7):2645-51. doi: 10.1523/JNEUROSCI.3501-13.2014. PMID 24523553
- [Background] Walker-Batson D, Curtis S, Natarajan R, Ford J, Dronkers N, Salmeron E, Lai J, Unwin DH. A double-blind, placebo-controlled study of the use of amphetamine in the treatment of aphasia. Stroke. 2001 Sep;32(9):2093-8. doi: 10.1161/hs0901.095720. PMID 11546902
- [Derived] Stockbridge MD, Fridriksson J, Sen S, Bonilha L, Hillis AE. Protocol for Escitalopram and Language Intervention for Subacute Aphasia (ELISA): A randomized, double blind, placebo-controlled trial. PLoS One. 2021 Dec 23;16(12):e0261474. doi: 10.1371/journal.pone.0261474. eCollection 2021. PMID 34941929